CLINICAL TRIAL: NCT02733900
Title: Study of Modifications of the Composition and Structure in the Aseptic Osteonecrosis of the Femoral Head and Etiopathogenic MRI Correlations
Brief Title: Modifications of the Subchondral Bone in Aseptic Osteonecrosis of the Femoral Head
Acronym: ONTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC-P0044
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Femur Head Necrosis
Keywords: aseptic osteonecrosis; femoral head; micro scanner; Raman spectrometry; MRI
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteonecrosis group (Experimental): Patients with an aseptic osteonecrosis of the femoral head
  Interventions: Procedure: femoral head removal
- Control group (Other): Patients with coxarthrosis
  Interventions: Procedure: femoral head removal

INTERVENTIONS:
Procedure: femoral head removal

SUMMARY:
In this study, the aim is to identify the modifications responsible for aseptic osteonecrosis of the femoral head and its structural evolution by the association of the micro scanner analysis and Raman spectrometry performed on the femoral heads removed during hip replacements. The study of femoral heads will allow the analysis of bone tissue at two different scales, both correlated with the biomechanical properties of the bone. Also, the association with preliminary MRI analysis will provide pathogenic explanations correlated to these modifications.

ELIGIBILITY:
Inclusion Criteria for experimental group:

* Men
* Patients aged from 25 to 70 years
* Patient with an aseptic osteonecrosis of the femoral head established by medical Imaging (CT-scan, MRI or radiography)
* FICAT stage 3 or 4
* osteonecrosis etiologies : alcohol, corticosteroid therapy, idiopathic
* Surgical indication of hip prosthesis determined

Inclusion Criteria for control group:

* Men
* Patients aged from 40 to 70 years
* Patient with a primitive coxarthrosis
* Surgical indication of hip prosthesis determined

Exclusion Criteria for the 2 groups:

* Other causes of osteonecrosis (coagulopathy, barotrauma, trauma)
* Prior fracture of the upper extremity of the femur
* Prior cancer and hematological malignancies with bone locations
* Prior debilitating bone diseases
* Patient refusal to participate in the study
* Patient who isn't affiliated to a social security regimen

Ages: 25 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Osseous modifications responsible of osteonecrosis | through the study completion, an average of 18 months

SECONDARY OUTCOMES:
Total cross-sectional area | through the study completion, an average of 27 months
  by using a contrast-enhanced nano-CT for the subchondral plate in necrotic zone, juxta-necrotic zone, remotely of the necrotic zone and cortical of the femoral collar
cortical bone area | through the study completion, an average of 27 months
  by using a contrast-enhanced nano-CT for the subchondral plate in necrotic zone, juxta-necrotic zone, remotely of the necrotic zone and cortical of the femoral collar
cortical area fraction | through the study completion, an average of 27 months
  by using a contrast-enhanced nano-CT for the subchondral plate in necrotic zone, juxta-necrotic zone, remotely of the necrotic zone and cortical of the femoral collar
cortical thickness | through the study completion, an average of 27 months
  by using a contrast-enhanced nano-CT for the subchondral plate in necrotic zone, juxta-necrotic zone, remotely of the necrotic zone and cortical of the femoral collar
bone volume fraction | through the study completion, an average of 27 months
  by using a contrast-enhanced nano-CT for the subchondral trabecular bone
trabecular number | through the study completion, an average of 27 months
  by using a contrast-enhanced nano-CT for the subchondral trabecular bone
trabecular separation | through the study completion, an average of 27 months
  by using a nano-CT for the subchondral trabecular bone
trabecular thickness | through the study completion, an average of 27 months
  by using a contrast-enhanced nano-CT for the subchondral trabecular bone
Physico-chemical composition of the trabecular subchondral bone | through the study completion, an average of 27 months
  mineralisation, carbonation, crystallinity, secondary structure of collagen, maturity of collagen, relative content of proteoglycans. These measures will be done for the trabecular subchondral bone in necrotic zone, juxta-necrotic zone, remotely of the necrotic zone and in the cortical of the femoral collar
Existence and extent of edema | through the study completion, an average of 27 months
  this measure will be done on the T2-weighted sequences with fat suppression
Perfusion MRI sequence | through the study completion, an average of 27 months
  morphological aspect of the enhancement curve, semi-quantitative parameters (slope, area under the curve, time to peak) and pharmacokinetic parameters
Medullary fat fraction in T1-weighted DIXON method | through the study completion, an average of 27 months
  border of osteosclerosis, identification of a necrotic zone, extent of this zone
Evaluation of osteocyte and adipocyte viability in hematoxylin-eosin-saffron (HES) staining | through the study completion, an average of 27 months
Number and ramifications of sub-chondral microvessels by immuno-labeling with CD21 | through the study completion, an average of 27 months
Evaluation of the number of osteoclasts by TRAP (tartrate acid Phosphatase) staining | through the study completion, an average of 27 months
Mankin score for cartilage degradation by Safranin O staining | through the study completion, an average of 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Pascart, MD, Principal Investigator — Hospital Group of the Catholic Institute of Lille
Locations (2):
- France (2):
  - Hospital Salengro CHU Lille, Lille
  - Hospital Group of the Catholic Institute of Lille, Lomme

IPD SHARING:
Plan to Share IPD: No